CLINICAL TRIAL: NCT01240850
Title: Medical Therapy in Idiopathic Retroperitoneal Fibrosis: a Multicenter, Randomized, Controlled Trial of Prednisone vs Low-dose Prednisone Plus Methotrexate
Brief Title: Methotrexate as a Steroid-sparing Agent in Idiopathic Retroperitoneal Fibrosis: a Randomised, Multicenter Trial
Acronym: FIPREDEX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Responsible Party: Prof Carlo Buzio, University of Parma
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: FARM79BKPY; 2008-007353-12 (EudraCT Number)
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Idiopathic Retroperitoneal Fibrosis; Perianeurysmal Retroperitoneal Fibrosis; Chronic Periaortitis
Keywords: Retroperitoneal fibrosis; Inflammatory aneurysms; Methotrexate; Prednisone; Aorta
MeSH Terms: conditions — Retroperitoneal Fibrosis | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone (Active Comparator)
  Interventions: Drug: Prednisone
- Methotrexate+Prednisone (Experimental)
  Interventions: Drug: Methotrexate+Prednisone

INTERVENTIONS:
Drug: Methotrexate+Prednisone — Methotrexate will be added at a dose of 0.3 mg/kg/week (maximum dose, 20 mg/week, orally) to a reduced-dose prednisone regimen
  Arms: Methotrexate+Prednisone
Drug: Prednisone
  Arms: Prednisone

SUMMARY:
Chronic periaortitis is a clinico-pathological entity encompassing idiopathic retroperitoneal fibrosis and perianeurysmal retroperitoneal fibrosis. The treatment of this disease is generally based on the use of glucocorticoids, which are often effective. However, prolonged steroid treatments are usually needed to achieve a sustained remission; additionally, patients frequently develop disease relapses following treatment discontinuation, therefore they may be exposed to high cumulative doses of glucocorticoids.

Preliminary data reported in the literature show that methotrexate may be effective in combination with prednisone for retroperitoneal fibrosis. In addition, methotrexate is often used as a steroid-sparing agent in different inflammatory diseases.

The aim of this study is to evaluate whether a treatment with low-dose prednisone plus methotrexate is non-inferior to conventional dose-prednisone in achieving remission in retroperitoneal fibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of idiopathic retroperitoneal fibrosis or chronic periaortitis; written informed consent

Exclusion Criteria:

* Secondary forms of retroperitoneal fibrosis (e.g. drugs, surgery, neoplasms, infections)
* Previous medical therapy for retroperitoneal fibrosis
* Renal failure with creatinine >2 mg/dl which proved not to be reversible after ureteral decompression
* Hypersensitivity to the study drugs
* Pregnancy
* Active infections or malignant neoplasms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-05; Primary Completion 2012-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Remission rate by the end of treatment

SECONDARY OUTCOMES:
Reduction in size of the retroperitoneal mass on CT/MRI scans
Rate of post-treatment relapses
Treatment-related toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Vaglio, MD, PhD, Principal Investigator — Parma University Hospital
Locations (1):
- Nephrology Unit, University Hospital of Parma, Parma, Parma, Italy

REFERENCES:
- [Background] van Bommel EF, Siemes C, Hak LE, van der Veer SJ, Hendriksz TR. Long-term renal and patient outcome in idiopathic retroperitoneal fibrosis treated with prednisone. Am J Kidney Dis. 2007 May;49(5):615-25. doi: 10.1053/j.ajkd.2007.02.268. PMID 17472843
- [Background] Vaglio A, Palmisano A, Corradi D, Salvarani C, Buzio C. Retroperitoneal fibrosis: evolving concepts. Rheum Dis Clin North Am. 2007 Nov;33(4):803-17, vi-vii. doi: 10.1016/j.rdc.2007.07.013. PMID 18037118
- [Background] Vaglio A, Salvarani C, Buzio C. Retroperitoneal fibrosis. Lancet. 2006 Jan 21;367(9506):241-51. doi: 10.1016/S0140-6736(06)68035-5. PMID 16427494
- [Background] Warnatz K, Keskin AG, Uhl M, Scholz C, Katzenwadel A, Vaith P, Peter HH, Walker UA. Immunosuppressive treatment of chronic periaortitis: a retrospective study of 20 patients with chronic periaortitis and a review of the literature. Ann Rheum Dis. 2005 Jun;64(6):828-33. doi: 10.1136/ard.2004.029793. PMID 15897305
- [Derived] Peyronel F, Palmisano A, Maritati F, Alberici F, Urban ML, Gianfreda D, Rossi GM, Fenaroli P, Bettiol A, Moroni G, Vaglio A. Methotrexate and low-dose prednisone in idiopathic retroperitoneal fibrosis: a randomised clinical trial. J Autoimmun. 2025 Dec;157:103487. doi: 10.1016/j.jaut.2025.103487. Epub 2025 Sep 19. PMID 40974866